CLINICAL TRIAL: NCT04172324
Title: The Effect of a Novel Gait Trainer, the Hibbot, on the Development of Crouch Gait in Children With Cerebral Palsy
Brief Title: Walking in the HIBBOT: is Gait Improved?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Ann Hallemans, Assistent Professor, Research Group MOVANT, Department of Rehabilitation Sciences and Physiotherapy - Head of the Multidisciplinary Motor Center Antwerp, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18/44/509
Record Dates: First submitted 2019-11-18; First posted 2019-11-21 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Cerebral Palsy
Keywords: gait; biomechanics
MeSH Terms: conditions — Cerebral Palsy | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hibbot (Experimental)
  Interventions: Device: HIBBOT; Other: Standard Care
- Standard Care (Active Comparator)
  Interventions: Other: Standard Care

INTERVENTIONS:
Device: HIBBOT — Hibbot is an assistive mechanical device, lightweight and portable. The mechanism of the Hibbot manages to control all degrees of freedom (3x rotation and 3x translation) at the level of the pelvis and lower trunk. The goal is to maximize a child's own muscle activity and postural control while giving as minimal support as needed.
  Arms: Hibbot
Other: Standard Care — Standard care involves the standard physiotherapy the child would get during clinical care.

SUMMARY:
The aim of the study is to assess the impact of the innovative walking aid HIBBOT on the functions, activity and participation of young children with Cerebral Palsy, in comparison with conventional walking aids.

ELIGIBILITY:
Inclusion Criteria:

* At risk of or diagnosed with cerebral palsy, based on MRI (uCP 86 - 89 % sensitivity) or HINE (uCP 98% ) or standard motor assessment
* age 18 months - 6 years
* GMFCS level II - IV =with potential (=able to stand and walk when supported by a therapist at the level of the pelvis and lower trunk)
* Sufficient cooperation to complete the tests.

Exclusion Criteria:

* Hip dysplasia
* Fixed contractures in the lower limb
* Botox infiltration < 6 months prior to inclusion
* Surgery < 12 months prior to inclusion
* Insufficient understanding of the interventon and tests (based on mental level assessment)
* Refractary epilepsia

Ages: 18 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Lower limb kinematics during walking in degrees | baseline (at intake, T0) and after the intervention period (3 months, T1)
  The gait pattern is assessed by instrumented 3D gait analysis. Joint rotation angles of the major joints of the lower limbs will be described during walking.
Change in Muscle activation patterns during gait in microvolts | baseline (at intake, T0) and after the intervention period (3 months, T1)
  Surface electromyography signals will be recorded during gait

SECONDARY OUTCOMES:
Lower limb kinematics during walking in degrees | at follow up (12 months after intake, T2)
  The gait pattern is assessed by instrumented 3D gait analysis. Joint rotation angles of the major joints of the lower limbs will be described during walking.
Muscle activation patterns during gait in microvolts | at follow up (12 months after intake, T2)
  Surface electromyography signals will be recorded during gait

CONTACTS AND LOCATIONS:
Locations (1):
- University of Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Analytic Code
Time Frame: At finalisation of the study and for a period of 5 years
Access Criteria: The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.